CLINICAL TRIAL: NCT05244330
Title: Effectiveness of COVID-19 Vaccines Against the SARS-COV-2 Delta (B.1.617.2) in China-A Real World Study
Brief Title: Effectiveness of COVID-19 Vaccines Against the SARS-COV-2 Delta (B.1.617.2)
Acronym: FASTER
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2022LSK-001
Record Dates: First submitted 2022-01-13; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-01

CONDITIONS: SARS CoV 2 Infection
Keywords: SARS-COV-2 Delta (B.1.617.2 ); vaccine; China; protective effect
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Partial vaccination: One dose of vaccine received at least 7 days prior to study enrollment
- Full vaccination: Two doses of COVID-19 vaccine received at least 7 days prior to study enrollment
- Unvaccinated: No dose of COVID-19 vaccine for at least 7 days prior to study enrollment

INTERVENTIONS:
Other:

SUMMARY:
Up to now, Corona Virus Disease 2019 (COVID-19) continues to spread rapidly around the world. From the beginning of the epidemic to the present, severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has continuously evolved and mutated, producing transmissible and virulent variants. At present, the infection rate of Delta variant strains is still increasing globally. The epidemic strain of novel coronavirus infection in Xi 'an city is δ (B.1.617.2). SARS-CoV-2 Delta has more infectious, higher viral load and shorter incubation period than other SARS-COV-2 delta strains. Several studies have shown that the protective efficacy of vaccines against different SARS-COV-2 virus variants is different, and SARS-COV-2 viral load is closely related to transmission, clinical phenotype and prognosis of infected patients. According to the notice of Xi'an Municipal Health Commission, a total of 2,139 local confirmed cases were reported in Xi 'an on January 10,2022, and the proportion of severe cases was 2.36%, which was significantly lower than the 7% of nation since the second half of 2020. According to the preliminary investigation by the applicant's team, the severe illness rate in Xi'an has decreased significantly, which benefits from the active promotion of domestic vaccination, early intervention, and use of neutralizing antibodies. The purpose of this study is to analyze the effects of vaccination on nucleic acid turning negative, clinical characteristics and prognosis of patients infected with SARS-COV-2 delta, and to clarify the protective effects of vaccination, which is of great significance for the prevention and control of the SARS-COV-2 delta (B.1.617.2) in Xi' an.

DETAILED DESCRIPTION:
In this study, through follow-up of SARS-COV-2 Delta infection patients in Xi 'an, Shaanxi Province, China, exploring the effects of vaccination on nucleic acid turning negative, clinical characteristics and prognosis of patients infected with SARS-COV-2 Delta, so as to clarify the protective effects of vaccination on SARS-COV-2 Delta.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with SARS-COV-2 Delta infection
* Clear vaccination information
* Plasma viral load measurements within 24 hours of admission to the hospital
* Performing continuous plasma viral load measurements
* Obtaining informed consent

Exclusion Criteria:

* Pregnant women
* Clinical diagnosis of organ dysfunction or failure before infection
* Long-term use of immunosuppressants or immunodeficiency patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with SARS-COV-2 Delta infection in Xi'an, Shaanxi Province, China, from December 2021 to January 2022
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
the proportion of severe and critical cases | during hospitalization, an average of 1 month
  the proportion of severe and critical cases during hospitalization

SECONDARY OUTCOMES:
the duration of viral shedding | during hospitalization, an average of 1 month
  the duration of SARS-COV-2 Delta (B.1.617.2) shedding

CONTACTS AND LOCATIONS:
Overall Officials: Kai Qu, Doctor, Study Director — First Affiliated Hospital Xi'an Jiaotong University; Guoliang Li, Doctor, Study Director — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian JiaotongUniversity, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided